CLINICAL TRIAL: NCT05505825
Title: A Phase Ib/II Clinical Study of Anti-PD-1 and CTLA-4 Bispecific Antibody, Cadonilimab(AK104), in Combination With Chiauranib in the Treatment of Patients With Extensive Stage Small Cell Lung Cancer Who Failed First-line Platinum-based Chemotherapy in Combination With Programmed Cell Death-1(PD1)/Programmed Cell Death Protein Ligand-1(PDL1) Inhibitors
Brief Title: A Study of AK104 in Combination With Chiauranib in Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-212
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: SCLC,Extensive Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 once every 3 weeks and Chiauranib once a day (Experimental): Subjects receive AK104 once every 3 weeks plus Chiauranib once a day until intolerable toxicity, no more clinical benefit as judged by the investigator, or completion of 24 months of treatment, or meeting other criteria for termination of treatment in the protocol, whichever occurs first.
  Interventions: Drug: AK104 IV infusion；Chiauranib oral

INTERVENTIONS:
Drug: AK104 IV infusion；Chiauranib oral — AK104 IV infusion once every 3 weeks；Chiauranib once a day oral

SUMMARY:
A Phase Ib/II open label,international multicentre study to evaluate the efficacy and safety of anti-PD-1 and CTLA-4 bispecific antibody AK104 in combination with Chiauranib in Patients with Extensive Stage Small Cell Lung Cancer Who Failed First-line Platinum-based Chemotherapy in Combination with PD1/PDL1 Inhibitors

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) consists 15% of the lung cancer.Because of the high malignancy, poor cell differentiation, and rapid proliferation of SCLC, 65% of the patients were in the extensive stage at their first presentation in the hospital with a very poor prognosis. There were few options of second-line therapies for patients who experienced progress disease during or after the end of first-line platinum-based regimens. Several studies showed that PD-1/PD-L1 inhibitors had synergistic anti-tumor effects with anti-vascular endothelial growth factor(VEGF) agents, i.e., PD-1/PD-L1 inhibitors could restore the anti-tumor effect of the immune system by blocking PD-L1, and anti-VEGF agents could improve the efficacy of the former by blocking the immunosuppressive effect of VEGF and promoting the infiltration of T cells in tumor tissues. Immunotherapy in combination with antiangiogenic therapy may become a trend in the treatment of extensive stage small cell lung cancer(ES-SCLC). The aim of this international multicentre phase Ib/II trial is to evaluate the efficacy-objective response rate according to RECIST criteria and safety-incidence and severity of adverse events.The patients' recruitment timeframe is set at 16 months and approximately 42 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form (ICF) voluntarily.
2. Aged ≥ 18 to ≤ 75 years.
3. Eastern Cooperative Oncology Group(ECOG) performance status score of 0 or 1.
4. Life expectancy≥ 3 months.
5. Histologically or cytologically confirmed ES-SCLC according to the Veterans Administration Lung Study Group(VALG) stage.
6. Phase Ib and II: Subjects with ES-SCLC who have failed prior first-line platinum-based chemotherapy in combination with PD1/PDL1 inhibitors will be enrolled.
7. At least 1 measurable lesion per RECIST v1.1, which is applicable for repeated accurate measurement. Brain metastatic lesions are not considered target lesions.
8. Adequate organ function.
9. Women of childbearing potential must have a negative urine or serum pregnancy test
10. If a nonsterile male subject has sexual intercourse with a female partner of childbearing potential, he must use an effective method of contraception from the start of screening until Day 120 after the last dose; it should be discussed with the Investigator whether contraception should be discontinued after this time point.
11. Subjects must be willing and able to comply with the scheduled visits, treatment regimens, laboratory tests, and other requirements in the study.

Exclusion Criteria:

1. Malignancies other than SCLC within 3 years prior to enrollment. However, subjects with other malignancies that have been cured are eligible.
2. Concurrent enrollment in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study.
3. Subjects whose imaging at screening shows that the tumor encircles important blood vessels or has significant necrosis and cavitation, and the subjects'participation is associated with a risk of hemorrhage.
4. Tumor invasion of surrounding vital organs and blood vessels.
5. Subjects who had active autoimmune disease that required systemic treatment in the past two years.
6. Subjects with prior history of non-infectious pneumonitis/interstitial lung disease requiring systemic glucocorticoid therapy or with non-infectious pneumonitis at present.
7. Presence of metastases to brainstem, meninges and spinal cord, or spinal cord compression.
8. Subjects with pleural effusion, pericardial effusion, or ascites that are clinically symptomatic or require drainage.
9. Subjects with unresolved toxicity due to prior anti-tumor therapy, defined as failure to recover to National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE) v5.0 Grade 0 or 1 (except for alopecia) or to the levels specified in the inclusion/exclusion criteria.
10. Subjects who cannot swallow pills, and who have malabsorption syndrome, or any condition affecting gastrointestinal absorption. Subjects with active or prior history of definite inflammatory bowel disease.
11. Subjects with a history of immunodeficiency; a positive human immunodeficiency virus (HIV) antibody test; and current long-term use of systemic corticosteroids or other immunosuppressants.
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Subjects who had major surgical procedure or serious trauma within 30 days prior to the first dose, or a major scheduled surgery within 30 days after the first dose; subjects who had minor local surgery within 3 days prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  ORR is proportion of subjects with complete response(CR) or partial response(PR), based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1
Incidence and severity of adverse events(AEs) | Up to approximately 2 years
  Incidence and severity of AEs is aim to evaluate the safety of AK104 in combination with Chiauranib.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  Disease control rate (DCR) is defined as the proportion of subjects achieving a best of response(BOR) of confirmed CR and PR and stable disease(SD) per RECIST v1.1.
duration of response (DoR) | Up to approximately 2 years
  Duration of response (DoR) is defined as the period from the first documentation of confirmed response (CR or PR) to the first documentation of progressive disease(PD) (as per RECIST v1.1) or death due to any cause, whichever occurs first.
time to response (TTR) | Up to approximately 2 years
  Time to response (TTR) is defined as the time from the first dose of investigational products until the first confirmation of CR or PR.
progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) is defined as the time from the first dose of investigational products until documentation of PD (as per RECIST v1.1) or death due to any cause, whichever occurs first.
overall survival (OS) | Up to approximately 2 years
  Overall survival (OS) is defined as the time from the first dose of investigational products until death due to any cause.
Pharmacokinetics(PK) profiles | Up to approximately 2 years
  Serum concentrations of AK104 and plasma concentrations of Chiauranib in individual subjects at different time points after administration of AK104 in combination with Chiauranib.
Immunogenicity assessment | Up to approximately 2 years
  The immunogenic potential of AK104 in combination with Chiauranib will be assessed by summarizing the number and percentage of subjects with detectable antidrug antibody(ADA).

OTHER OUTCOMES:
alpha thalassemia/mental retardation X-linked(ATRX) gene mutation status | Up to approximately 2 years
  The ATRX gene mutation status in peripheral blood will be determined, and its correlation with efficacy indicators such as ORR, PFS and OS will be analyzed.
SCLC subtype | Up to approximately 2 years
  The expression of proteins related to SCLC subtype in tumor tissue samples will be detected by immunohistochemistry (IHC) and its correlation with efficacy will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Professor, Principal Investigator — Jilin Province Cancer Hospital
Locations (7):
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Jilin Province Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No